CLINICAL TRIAL: NCT05881369
Title: Exploring the Clinical Trial Journey of Patients in Substance Abuse Disorder Clinical Trials
Brief Title: Examining Clinical Research Participation for Substance Abuse Disorder Patient
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 91257336
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Substance Abuse Disorder
Keywords: substance abuse disorder
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical study participation percentages haven't always been fully representative of a given demographic.

The goal is to find out which aspects of a clinical trial may make it more difficult for patients to take part or see it through.

The data will be evaluated through different demographic lenses and identify trends that could help improve the experience of future substance abuse disorder patients during clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
* Participant has a diagnosis of substance abuse disorder.
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.

Exclusion Criteria:

* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
* Pregnant or lactating woman
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or interfere with the interpretation of safety results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Substance abuse disorder patients who are actively considering involvement in an observational clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a substance abuse disorder clinical study. | 3 months
Number of substance abuse disorder patients who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kock P, Froelich K, Walter M, Lang U, Dursteler KM. A systematic literature review of clinical trials and therapeutic applications of ibogaine. J Subst Abuse Treat. 2022 Jul;138:108717. doi: 10.1016/j.jsat.2021.108717. Epub 2021 Dec 30. PMID 35012793
- [Background] Jaguga F, Kwobah E. A review of the public sector substance use disorder treatment and prevention systems in Kenya. Subst Abuse Treat Prev Policy. 2020 Jul 20;15(1):47. doi: 10.1186/s13011-020-00291-5. PMID 32690036
- [Background] Tull MT, Gratz KL. The impact of borderline personality disorder on residential substance abuse treatment dropout among men. Drug Alcohol Depend. 2012 Feb 1;121(1-2):97-102. doi: 10.1016/j.drugalcdep.2011.08.014. Epub 2011 Sep 9. PMID 21907503

DOCUMENTS (1):
  • Informed Consent Form (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT05881369/ICF_000.pdf